CLINICAL TRIAL: NCT02218411
Title: Effectiveness of a Video-supported Group-based Otago Exercise Programme on Physical Performance in Community-dwelling Older Adults: a Pilot Randomized Controlled Trial
Brief Title: Video-supported Group-based Otago Exercise Programme on Physical Performance in Older Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Eva Segura Ortí, Effectiveness of a video-supported group-based Otago exercise programme on physical performance in community-dwelling older adults: a pilot randomized controlled trial, Cardenal Herrera University
Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEU UCH
Record Dates: First submitted 2014-07-14; First posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Healthy Aging
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise (Experimental): Exercises routine based on the Otago exercise programme
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — Exercises routine based on the Otago exercise programme

SUMMARY:
The purpose of this study was to evaluate the effects of a video-supported group-based Otago exercise programme intervention on balance, mobility, physical performance and aerobic endurance in community-dwelling older adults 65+ years old.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years and older.
* Living in the community (Valencia, Spain).
* Able to ambulate independently without a walking aid.
* Have no severe medical contraindication for physical activity.
* Able to communicate.
* Have self-reported visual and auditory capacities to follow commands.
* Provide signed informed consent.

Exclusion Criteria:

* Unable to ambulate independently.
* Mini-mental state examination score of <24.
* Barthel Index score of <80.
* Severe visual and auditory disabilities.
* Unstable cardiovascular disease.
* Neurological disorder that could compromise them from exercising.
* Upper or lower extremity fracture in the past year.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-09; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in the Timed Up and Go test | Pre intervention and after 4-month intervention
  General mobility measurement

SECONDARY OUTCOMES:
Change in the Berg Balance Scale | Pre intervention and after 4-month intervention
  Functional Balance measurement
Change in the 6.min Walk Test | Pre intervention and after 4-month intervention
  Aerobic Endurance Measurement
Change in the One-Leg Stand | Pre intervention and after 4-month intervention
  One-leg Balance Measurement
Change in the Short Physical Performance Battery | Pre intervention and after 4-month intervention
  Lower Limb Functional Measurement

CONTACTS AND LOCATIONS:
Overall Officials: Vicent Benavent-Caballer, PT, MS, Principal Investigator — CEU UCH

REFERENCES:
- [Derived] Benavent-Caballer V, Rosado-Calatayud P, Segura-Orti E, Amer-Cuenca JJ, Lison JF. The effectiveness of a video-supported group-based Otago exercise programme on physical performance in community-dwelling older adults: a preliminary study. Physiotherapy. 2016 Sep;102(3):280-6. doi: 10.1016/j.physio.2015.08.002. Epub 2015 Sep 1. PMID 26395209